CLINICAL TRIAL: NCT04994808
Title: A Phase II Randomized Study to Assess Outcomes With Treosulfan-Based Versus Clofarabine-Based Conditioning in Patients With Myelodysplastic Syndromes With Excess Blasts (MDS-EB), or Acute Myeloid Leukemia (AML) Undergoing Allogeneic Hematopoietic Cell Transplantation (HCT)
Brief Title: Treosulfan-Based Versus Clofarabine-Based Conditioning Before Donor Hematopoietic Stem Cell Transplant for the Treatment of Myelodysplastic Syndromes or Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Medexus Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1121616; NCI-2021-07474 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10598 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Clofarabine; fludarabine; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Whole-Body Irradiation; treosulfan; Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (treosulfan, fludarabine, TBI, HCT) (Experimental): Patients receive treosulfan IV over 2 hours on days -6 to -4 and fludarabine IV over 30 minutes on days -6 to -2. Patients also undergo TBI followed by HCT on day 0. Patients undergo ECHO or MUGA and lumbar puncture pre-transplant and undergo bone marrow aspiration, bone marrow biopsy, and collection of blood samples at pre-transplant and post-transplant.
  Interventions: Drug: Fludarabine; Procedure: Hematopoietic Cell Transplantation; Radiation: Total-Body Irradiation; Drug: Treosulfan; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Procedure: Lumbar Puncture; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Biospecimen Collection
- Arm B (clofarabine, TBI, HCT) (Experimental): Patients receive clofarabine IV over 2 hours on days -6 to -2. Patients also undergo TBI followed by HCT on day 0. Patients undergo ECHO or MUGA and lumbar puncture pre-transplant and undergo bone marrow aspiration, bone marrow biopsy, and collection of blood samples at pre-transplant and post-transplant.
  Interventions: Drug: Clofarabine; Procedure: Hematopoietic Cell Transplantation; Radiation: Total-Body Irradiation; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Procedure: Lumbar Puncture; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Clofarabine — Given IV
  Other Names: Clofarex; Clolar
  Arms: Arm B (clofarabine, TBI, HCT)
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
  Arms: Arm A (treosulfan, fludarabine, TBI, HCT)
Procedure: Hematopoietic Cell Transplantation — Undergo HCT
  Other Names: HCT; Hematopoietic Stem Cell Infusion; Hematopoietic Stem Cell Transplantation; HSCT; Stem Cell Transplant; stem cell transplantation
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: SCT_TBI; TBI; Total Body Irradiation; Whole Body Irradiation; Whole-Body Irradiation
Drug: Treosulfan — Given IV
  Other Names: 1,2,3, 4-Butanetetrol, 1,4-dimethanesulfonate, [R-(R*,S*)]-; Dihydroxybusulfan; Ovastat; Trecondi; Treosulphan; Tresulfon; Grafapex
  Arms: Arm A (treosulfan, fludarabine, TBI, HCT)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: MUGA; MUGA Scan; Multi-Gated Acquisition Scan
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; spinal tap
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection

SUMMARY:
This phase II trials studies the effect of treosulfan-based versus clofarabine-based conditioning regimens before donor hematopoietic stem cell transplant in treating patients with myelodysplastic syndromes or acute myeloid leukemia. Chemotherapy drugs, such as treosulfan, fludarabine, and clofarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy and total-body irradiation before a donor hematopoietic stem cell transplant helps kill cancer cells in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. When the healthy stem cells from a donor are infused into a patient, they may help the patient's bone marrow make more healthy cells and platelets and may help destroy any remaining cancer cells. This study may help doctors determine whether treosulfan-based or clofarabine-based conditioning regimen works better before donor hematopoietic stem cell transplant in treating patients with myelodysplastic syndromes or acute myeloid leukemia.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive treosulfan intravenously (IV) over 2 hours on days -6 to -4 and fludarabine IV over 30 minutes on days -6 to -2. Patients also undergo total-body irradiation (TBI) followed by HCT on day 0. Patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) and lumbar puncture pre-transplant and undergo bone marrow aspiration, bone marrow biopsy, and collection of blood samples at pre-transplant and post-transplant.

ARM B: Patients receive clofarabine IV over 2 hours on days -6 to -2. Patients also undergo TBI followed by HCT on day 0. Patients undergo ECHO or MUGA and lumbar puncture pre-transplant and undergo bone marrow aspiration, bone marrow biopsy, and collection of blood samples at pre-transplant and post-transplant.

After completion of study intervention, patients are followed up at days 28, 56, 84 and 180, years 1 and 1.5 and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years and =< 75 years
* Diagnosis of MDS-EB or AML: must have < 5% marrow blasts (by morphology and/or flow cytometry) at time of transplant
* Karnofsky performance score (KPS) >= 60% on pre-HCT evaluation
* Able to give informed consent
* Patients with previous autologous or allogeneic HCT may enroll
* DONOR: Human leukocyte antigen (HLA)-identical related donors or unrelated donors matched for HLA-A, B, C, DRB1, and DQB1 as defined by high resolution deoxyribonucleic acid (DNA) typing; mismatch for only one HLA allele at class I is allowed
* DONOR: Donors able to undergo peripheral blood stem cell collection. Only granulocyte colony-stimulating factor (G-CSF) mobilized peripheral blood stem cell (PBSC) will be permitted as an hematopoietic stem cell (HSC) source on this protocol

Exclusion Criteria:

* Presence of circulating blasts (in the blood) detected by standard pathology for patients with AML
* Presence of >= 5% circulating leukemic blasts (in the blood) detected by standard pathology for patients with MDS-EB
* Patients with promyelocytic AML
* Organ dysfunction

  * Cardiac: Ejection fraction < 35% (or, if unable to obtain ejection fraction, shortening fraction of < 26%) or cardiac insufficiency requiring treatment or symptomatic coronary artery disease. Patients with a shortening fraction < 26% may be enrolled if approved by a cardiologist
  * Pulmonary:

    * Diffusion capacity of the lung for carbon monoxide (DLCO) < 40%, total lung capacity (TLC) < 40%, forced expiratory volume in 1 second (FEV1) < 40% and/or receiving supplementary continuous oxygen. When pulmonary function test (PFT)s cannot be obtained, the 6-minute walk test (6 minute walk functional test [6MWT], also known as exercise oximetry) will be used: Any patient with oxygen saturation on room air of < 89% during a 6MWT will be excluded
    * The principal investigator (PI) must approve enrollment of all patients with pulmonary nodules
  * Renal: Serum creatinine should be within normal limits as specified by Standard Practice guidelines. For subjects with serum creatinine > upper limit of normal, a 24-hour creatinine clearance will be performed and should be equal to or more than the lower limit of normal
  * Hepatic: Patients with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension. Patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bridging fibrosis, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, or symptomatic biliary disease
* With active infectious disease requiring deferral of conditioning, as recommended by an infectious disease specialist
* Fungal infections with radiological progression after receipt of amphotericin B or active triazole for greater than 1 month
* With human immunodeficiency virus (HIV)-positivity or active infectious hepatitis because of possible risk of lethal infection when treated with immunosuppressive therapy
* With central nervous system (CNS) leukemia at the time of treatment
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers) or those with non-hematologic malignancies (except non-melanoma skin cancers) who have been rendered with no evidence of disease but have a greater than 20% chance of having disease recurrence within five years. This exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* With life expectancy severely limited by diseases other than malignancy
* Fertile men and women unwilling to used contraceptive techniques during treatment and for 12 months following
* Women who are pregnant or lactating
* With known hypersensitivity to treosulfan, fludarabine, or clofarabine
* The use of non-Food and Drug Administration (FDA) approved investigational drugs would not be allowed within 4 weeks of the initiation of conditioning (day -6 for both arms)
* Unable to give informed consent
* Patients suitable for and willing to receive a standard high intensity preparative regimen
* DONOR: Donor (or centers) who will exclusively donate marrow
* DONOR: Donors who are HIV-positive and/or, medical conditions that would result in increased risk for G-CSF mobilization and harvest of PBSC
* DONOR: Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment. This determination is based on the standard practice of the individual institution. The recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain a panel reactive antibody (PRA) screens to class I and class II antigens for all patients before HCT. If the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained. The donor should be excluded if any of the cytotoxic cross match assays are positive. For those patients with an HLA Class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results. A positive anti-donor cytotoxic cross match is an absolute donor exclusion
* DONOR: Donor is excluded if a patient is homozygous in the graft-rejection vector against the donor's mismatched HLA class I allele

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2026-01-22 (Actual); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | At 6 months after transplant

SECONDARY OUTCOMES:
Overall survival | At 1 year after transplant
Rate of non-relapse mortality | At 1 year after transplant
Relapse rate | At 1 year after transplant
Incidence of acute graft versus host disease | At 1 year after transplant
Duration of hospitalization | Up to day 100 post hematopoietic stem cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Phuong Vo, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT04994808/ICF_000.pdf